CLINICAL TRIAL: NCT06541249
Title: MethoTRExATE in MyelOpRolifErative Neoplasms (TREATMORE) Trial
Acronym: TREATMORE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, John Mascarenhas, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00071
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Polycythemia Vera (PV); Essential Thrombocythemia (ET); Myelofibrosis (MF)
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: Stage 1: 9 participants will be accrued to each of three cohorts of patients with MPNs: PV, ET, and MF. Low-dose, weekly MTX will be added to current therapy. If 0 responses occur within a given cohort, the study will be stopped within that cohort for futility; if ≥3 responses occur within a given cohort, the study will be stopped for early evidence of efficacy within that cohort.
  If 1-2 responses occur within any given cohort, that cohort will proceed to Stage 2. An additional 1 participant will be accrued to account for potential dropout. Stage 2: 9 additional participants will be accrued to each of three cohorts. If a total of >3 of 20 participants enrolled achieve responses in any cohort, the study will be considered successful and MTX worthy of further study within that cohort. An additional 1 participant will be accrued to account for potential dropout.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Myelofibrosis (MF) (Experimental): 18 patients with MF will be enrolled
  Interventions: Drug: Methotrexate (MTX)
- Polycythemia vera (PV) (Experimental): 18 patients with MF will be enrolled
  Interventions: Drug: Methotrexate (MTX)
- Essential thrombocythemia (ET) (Experimental): 18 patients with MF will be enrolled
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Methotrexate (MTX) — MTX has recently been identified as a dose-dependent JAK/STAT pathway inhibitor. 15mg will be given once a week orally.

SUMMARY:
Low-dose MTX is a widely used, inexpensive, and safe therapy used for decades and is well tolerated by patients with rheumatologic diseases. Recently, it was identified as a type 2 JAK inhibitor. If MTX proves to be safe and tolerable with a signal of clinical activity, this could have a significant benefit to patients with MPNs. Beyond the potential benefit of adding a type 2 JAK inhibitor to current therapy, this could signal the need to study MTX in MPNs further as a monotherapy. Discovering MTX as safe and clinically effective in MPNs could be profound on both a public health and global health scale for patients who are uninsured and cannot afford more expensive novel JAK inhibitors, or for those in countries where JAK inhibitors are not available. Accordingly, the research team deems it reasonable and prudent to assess the safety and efficacy of MTX in addition to current therapy for patients with MPN. The research team will evaluate patients for spleen responses, symptom responses, and cytologic responses. Correlative data will evaluate pharmacokinetic and disease modifying activity of MTX in MPNs to inform future clinical trials.

ELIGIBILITY:
Inclusion Criteria

* Be ≥18 years of age at time of signing the informed consent form (ICF)
* Must voluntarily sign ICF and be willing and able to adhere to the study visit schedule and all protocol requirements
* Have a pathologically confirmed diagnosis of PV, ET, PMF, post-ET-MF, or post-PV-MF as per WHO diagnostic criteria
* Participants with MF may have low, intermediate 1, intermediate 2, or high-risk disease by Dynamic International Prognostic Scoring System (DIPSS). Participants with PV and ET with both low- and high-risk disease may be included.
* Must have received at least 12 weeks of current MPN therapy at stable doses and have persistent clinical burden and/or cytologic abnormalities as defined by the following:

  * Clinical burden is defined as MPN-SAF TSS >12 points and/or palpable spleen of ≥5cm
  * Cytologic abnormalities include the following for each disease state:

    * MF:

      * Persistent leukocytosis as defined by WBC >12 x 109/L
    * PV:

      * Persistent therapeutic phlebotomy dependence (>2 phlebotomies within 24 weeks of screening, and >1 phlebotomy within 16 weeks of screening, as defined in the PROUD-PV studies) for a goal HCT <45% and/or
      * Leukocytosis as defined by WBC >12 x 109/L and/or
      * Thrombocytosis defined as platelet count >500 x 109/L
    * ET:

      * Persistent leukocytosis as defined by WBC >12 x 109/L and/or
      * Thrombocytosis defined as platelet count >500 x 109/L
  * Permitted concurrent MPN therapies include: aspirin, hydroxyurea, anagrelide, ropeginterferon alfa-2b, peginterferon alfa-2a, erythropoiesis-stimulating agents, phlebotomy, and/or ruxolitinib.

    * A stable dose is defined as 12 weeks of treatment without a change in dosing
    * Patients with myelofibrosis must be on stable dose of ruxolitinib
* Must have adequate organ function as demonstrated by the following:

  * AST, ALT <3x upper limit of normal (ULN) and no known history of cirrhosis
  * Total bilirubin <3mg/dL
  * Creatinine clearance (CrCl) >40 mL/min as estimated with the Cockcroft-Gault equation
  * Baseline platelet count >50 x 109/L for MF and >150 x 109/L for ET/PV
  * Baseline absolute neutrophil count (ANC) >1000
  * Peripheral blood blast count <10%
* ECOG performance status ≤2
* Life expectancy of at least six months
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and Cycle 1 Day 1 and must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * Recommended methods of birth control are:

    * The consistent use of an approved hormonal contraception (birth control pill/patches, rings), an intrauterine device (IUD), contraceptive injection (Depo-Provera), double barrier methods (diaphragm with spermicidal gel or condoms with contraceptive foam), sexual abstinence (no sexual intercourse), or sterilization
  * A woman of childbearing potential is any woman (regardless of sexual orientation, having undergone a tubal litigation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months
* Male participants must agree to use an adequate method of contraception and must not father a child or donate sperm starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Prescribed MTX for another indication
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months
* Have other invasive malignancies within the last 3 years, except non-melanoma skin cancer and localized, cured prostate and cervical cancer
* Have moderate or severe cardiovascular disease as defined by the following:

  * Have cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension
  * Have documented major ECG abnormalities (not responding to medical treatments)
* Be an organ transplant recipient other than bone marrow transplant
* Presence of active serious infection
* Have a known history B, or untreated hepatitis C infection
* Have a known history of pulmonary fibrosis, interstitial pneumonitis
* Have a known history of chronic pericardial effusions, pleural effusions, or ascites
* Have a known history of cirrhosis, or current heavy alcohol consumption
* Have impairment of gastrointestinal function or gastrointestinal disease that could significantly alter the absorption of MTX, including any unresolved nausea, vomiting, or diarrhea > CTCAE v5.0 grade 1
* Have known history of tuberculosis or severe fungal infection
* Is receiving specific concomitant medications that are contraindicated with MTX.
* Women who are pregnant or lactating, or plan to become pregnant during trial period
* Have any serious, unstable medical or psychiatric condition that would prevent (as judged by the Investigator) the participant from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MF Overall response rate | at 24 weeks
  MF overall response rate, defined as Clinical Improvement (CI) or greater per the IWG-MRT and ELN Response Criteria for MF (2013).
  CI or greater is defined as changes in the spleen, hemoglobin, and symptoms.
PV and ET Overall response rate | at 24 weeks
  PV overall response rate, defined as complete response (CR) or partial response (PR) by modified 2013 ELN criteria. CR response is defined as a lasting reduction in spleen size, symptom improvement, a reduction in platelet and white cell count. As well as changes in bone marrow biopsy.
  PR response is defined as lasting reduction in spleen size, symptom improvement, a reduction in platelet and white cell count.

SECONDARY OUTCOMES:
Adverse event Grade | Up to 48 Weeks
  The safety and the tolerability of treatment will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. This standardized system grades adverse events on a scale from 1 (mild) to 5 (death). Higher grades indicate more severe adverse events, with lower grades and fewer events suggesting better safety of the treatment.
Number of Participants with Myeloproliferative Neoplasm Symptom Assessment Form Score >50% | Up to 48 Weeks
  Symptom improvement response is defined as a number of participants with improvement in symptoms response as defined by Myeloproliferative Neoplasms Symptoms Assessment Form (MPN-SAF). The MPN-SAF is a questionnaire that measures certain symptoms and how they improve throughout the study, from baseline. The questionnaire is divided into 4 sections - 1: 16 questions about the most common symptoms in these disease types, rated from 0 (lowest impact) to 10 (biggest impact); 2: Highest grade of fever; 3: Unintentional weight loss; 4. Quality of life, rated from 0 (as good as it can be) to 10 (as bad as it can be).
Spleen Response Rate | Up to 48 Weeks
  Spleen response rate, defined as baseline splenomegaly palpable at 5-10cm becomes not palpable, or baseline splenomegaly of >10cm decreases by >50% by palpation.
Anemia Response Rate | Up to 48 Weeks
  Anemia response rate will be measured as clinical improvement if patient hemoglobin increase by 2g/dl from baseline and/or become transfusion independent, according to International Working Group for Myelofibrosis Research and Treatment IWG-MRT criteria (MF cohort).
Change in baseline hematocrit (PV cohort) | Baseline and 48 Weeks
  The change in the proportion of red blood cells in the blood measured using a hematocrit test. A hematocrit test measures the volume of packed red blood cells relative to whole blood. This is represented as a ratio. Change in baseline hematocrit will be measured for the PV cohort.
Change in baseline platelet count (ET cohort) | Baseline and 48 Weeks
  A platelet count is a lab test that measures how many platelets are in the blood. Platelets are particles in the blood that help the blood clot. Platelets may be counted to monitor or diagnose diseases, or to look for the cause of too much bleeding or clotting. Change in baseline platelet count will be measured for ET cohort.
Change from baseline monthly phlebotomy rate (PV cohort) | Baseline and 6 months
  Change in number of therapeutic phlebotomy over a 6 month period prior to starting the clinical trial compared to when the patient completes the clinical trial.
Change from baseline platelet transfusion dependence | Baseline and 48 Weeks
  Change in number of platelet transfusion over a 12 week period prior to starting the clinical trial compared to when the patient completes the clinical trial. (MF cohort)
Change from baseline pRBC transfusion dependence | at 24 and 48 Weeks
  Change in number of pRBC transfusion over a 12 week period prior to starting the clinical trial compared to when the patient completes the clinical trial. (MF cohort)
Change from baseline in dosing of cytoreductive agents (PV and ET Cohort) | Baseline and 48 Weeks
  Change from baseline in dosing of cytoreductive agents other than Methotrexate for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Ruttenberg Treatment Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices.)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to john.mascarenhas@mssm.edu. To gain access, data requestors will need to sign a data access agreement.